CLINICAL TRIAL: NCT00123903
Title: A Randomized, Double-blind, Positive-Controlled, Multicenter Study Comparing the Efficacy of Carvedilol Phosphate Modified Release Formulation (COREG MR) and Metoprolol Succinate Extended Release (TOPROL-XL) on the Reduction of Microalbuminuria in Patients With Hypertension and Microalbuminuria
Brief Title: COREG MR Versus TOPROL-XL On Reduction Of Microalbuminuria In Patients With Hypertension And Microalbuminuria
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: COR103560
Record Dates: First submitted 2005-07-22; First posted 2005-07-26 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Heart Failure, Congestive and Microalbuminuria
Keywords: hypertension; urine albumin:creatinine ratio; microalbuminuria
MeSH Terms: conditions — Heart Failure; Hypertension | interventions — Metoprolol; Lisinopril

INTERVENTIONS:
Drug: metoprolol xl
Drug: carvedilol MR
Drug: lisinopril
  Other Names: carvedilol MR; metoprolol xl

SUMMARY:
This study was designed to determine whether COREG MR is more effective than TOPROL-XL in reducing microalbuminuria in type 2 diabetic or non-diabetic patients with high blood pressure and microalbuminuria.

ELIGIBILITY:
Inclusion criteria:

* Documented history of hypertension.
* Must have been taking an ACE (angiotensin converting enzyme) inhibitor either alone or as part of an antihypertensive regimen for at least 8 weeks.
* Persistent microalbuminuria.

Exclusion criteria:

* History of heart attack, stroke, congestive heart failure, arrhythmia, type 1 or uncontrolled type 2 diabetes mellitus, liver or renal disease.
* Has been taking any non-ocular beta-blockers for any indication within three months prior to Pre-screening.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1220
Dates: Start 2005-07; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in urine albumin: creatinine ratio (ACR) at six months of maintenance therapy. | Baseline (Randomization Visit) and Month 6

SECONDARY OUTCOMES:
Percentage of participants who achieved normoalbuminuria at 6 months of maintenance therapy. | Month 6
Percentage of participants who progressed to macroalbuminuria after 6 months of maintenance therapy. | Month 6
Change from baseline to month 6 LOCF in High-sensitivity C-reactive protein (hs-CRP) | Baseline (Randomization Visit) and Month 6
Change from Pre-screening visit to month 6 LOCF in urine ACR. | Pre-screening Visit and Month 6
Change from baseline to visit to month 6 LOCF in lipids including total cholesterol, low density lipid (LDL), high density lipid (HDL) and Triglycerides (TG) | Baseline (Randomization visit) and Month 6
Changes from baseline in blood pressure (systolic and diastolic) at month 6 of treatment. | Baseline (Randomization Visit) and Month 6
Changes from baseline in heart rate at month 6 of treatment. | Baseline (Randomization visit) and Month 6
Percentage of participants who required add-on therapy to reach target blood pressure at any time during the study. | Up to 6 months
Number of participants with clinical chemistry parameters and hematology parameters of potential clinical concern at any time on-treatment. | Up to 6 months
Number of participants with vital signs of potential clinical concern at any time on-treatment. | Up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (84):
- United States (63):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Mobile, Alabama
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Fullerton, California
  - GSK Investigational Site, Inglewood, California
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Mission Viejo, California
  - GSK Investigational Site, Oakland, California
  - GSK Investigational Site, Redondo Beach, California
  - GSK Investigational Site, Colorado Springs, Colorado
  - GSK Investigational Site, Hollywood, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Pembroke Pines, Florida
  - GSK Investigational Site, Sarasota, Florida
  - GSK Investigational Site, Tampa, Florida
  - GSK Investigational Site, Decatur, Georgia
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Melrose Park, Illinois
  - GSK Investigational Site, Avon, Indiana
  - GSK Investigational Site, Elkhart, Indiana
  - GSK Investigational Site, Evansville, Indiana
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, Lafayette, Louisiana
  - GSK Investigational Site, Ayer, Massachusetts
  - GSK Investigational Site, Worcester, Massachusetts
  - GSK Investigational Site, Las Vegas, Nevada
  - GSK Investigational Site, Voorhees Township, New Jersey
  - GSK Investigational Site, Buffalo, New York
  - GSK Investigational Site, Camillus, New York
  - GSK Investigational Site, East Syracuse, New York
  - GSK Investigational Site, Kingston, New York
  - GSK Investigational Site, Port Chester, New York
  - GSK Investigational Site, Rochester, New York
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Greensboro, North Carolina
  - GSK Investigational Site, Raleigh, North Carolina
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Columbus, Ohio
  - GSK Investigational Site, Kettering, Ohio
  - GSK Investigational Site, Oklahoma City, Oklahoma
  - GSK Investigational Site, Oregon City, Oregon
  - GSK Investigational Site, Beaver, Pennsylvania
  - GSK Investigational Site, Havertown, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Reading, Pennsylvania
  - GSK Investigational Site, West Grove, Pennsylvania
  - GSK Investigational Site, East Providence, Rhode Island
  - GSK Investigational Site, Greer, South Carolina
  - GSK Investigational Site, Orangeburg, South Carolina
  - GSK Investigational Site, Johnson City, Tennessee
  - GSK Investigational Site, Beaumont, Texas
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Fort Worth, Texas
  - GSK Investigational Site, Galveston, Texas
  - GSK Investigational Site, Houston, Texas
  - GSK Investigational Site, Midland, Texas
  - GSK Investigational Site, San Antonio, Texas
  - GSK Investigational Site, Burke, Virginia
  - GSK Investigational Site, Springfield, Virginia
  - GSK Investigational Site, Edmonds, Washington
  - GSK Investigational Site, Olympia, Washington
  - GSK Investigational Site, Spokane, Washington
  - GSK Investigational Site, Wenatchee, Washington
- Canada (19):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, New Westminster, British Columbia
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Winnipeg, Manitoba
  - GSK Investigational Site, Bay Roberts, Newfoundland and Labrador
  - GSK Investigational Site, Brampton, Ontario
  - GSK Investigational Site, Hamilton, Ontario
  - GSK Investigational Site, Kitchener, Ontario
  - GSK Investigational Site, London, Ontario
  - GSK Investigational Site, Stoney Creek, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Charlottetown, Prince Edward Island
  - GSK Investigational Site, Montague, Prince Edward Island
  - GSK Investigational Site, Bonaventure, Quebec
  - GSK Investigational Site, Mirabel, Quebec
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Pointe-Claire, Quebec
  - GSK Investigational Site, Saint Romuald, Quebec
  - GSK Investigational Site, Trois-Rivières, Quebec
- Puerto Rico (2):
  - GSK Investigational Site, Río Grande, Puerto Rico
  - GSK Investigational Site, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: COR103560 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: COR103560 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: COR103560 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: COR103560 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: COR103560 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: COR103560 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: COR103560 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register